CLINICAL TRIAL: NCT01023334
Title: Combined Intracameral Lidocaine for Manual Small Incision Cataract Surgery Under Topical Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Wei Chen, Eye Hospital, Wenzhou Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10002
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2009-12

CONDITIONS: Cataract
Keywords: Topical analgesia; FlACC Pain Scale; intracameral lignocaine; Anesthetics; Physiological Effects of Drugs; Lidocaine
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraocular lidocaine,topical anesthesia,MSICS (Experimental): experimental group:manual small incision cataract surgery under topical anesthesia with intracameral lidocaine
  Interventions: Procedure: MSICS under topical anesthesia with intracameral lidocaine
- intracameral balanced salt solution,topical anesthesia,MSICS (Experimental): control group:manual small incision cataract surgery under topical anesthesia with intracameral balanced salt solution.
  Interventions: Procedure: MSICS under topical anesthesia with intracameral balanced salt solution.

INTERVENTIONS:
Procedure: MSICS under topical anesthesia with intracameral lidocaine — manual small incision cataract surgery(MSICS) under topical anesthesia with intracameral lidocaine
  Arms: Intraocular lidocaine,topical anesthesia,MSICS
Procedure: MSICS under topical anesthesia with intracameral balanced salt solution. — manual small incision cataract surgery(MSICS) under topical anesthesia with intracameral balanced salt solution.
  Arms: intracameral balanced salt solution,topical anesthesia,MSICS

SUMMARY:
The purpose of this study is to determine whether intraocular lidocaine increases patient comfort during the different stages of MSICS while under topical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women
* Cataract density grade III-V according to the Emery-Little system classification system
* Patients need to do manual small incision cataract surgery

Exclusion Criteria:

* Legal guardian(s) is/are not present for permission
* Any patient with a known sensitivity or allergy to Lidocaine or the "Caine" family of medicines.
* Patients with altered levels of pain perceptions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
observed levels of pain | one day

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, MD,PhD, Principal Investigator — Eye Hospital, Wenzhou Medical College, China
Locations (1):
- Eye Hospital, Wenzhou Medical College, Wenzhou, Zhejiang, China